CLINICAL TRIAL: NCT02454348
Title: NOrepinephrine and VasoprEssin Versus Norepinephrine aLone in Critically Ill Patients With Septic Shock (NOVEL Trial)
Brief Title: NOrepinephrine and VasoprEssin Versus Norepinephrine aLone in Critically Ill Patients With Septic Shock
Acronym: NOVEL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204265
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Shock, Septic
Keywords: septic shock; vasopressin; norepinephrine
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norepinephrine and vasopressin (Active Comparator): Norepinephrine (0.05 to 0.5 mcg/kg/min) and vasopressin (0.04 units/min) will be given by continuous infusion to achieve and maintain a target mean arterial pressure (65-75 mm Hg).
  Interventions: Drug: Vasopressin; Drug: Norepinephrine
- Norepinephrine (Active Comparator): Norepinephrine (0.05 to 0.5 mcg/kg/min) will be given by continuous infusion to achieve and maintain a target mean arterial pressure (65-75 mm Hg).
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Vasopressin — Subjects will receive vasopressin (0.04 units/min) by continuous infusion to achieve and maintain a target mean arterial pressure (65-75 mm Hg). The treating physician may choose the initial dosage of norepinephrine within the initial range of 0.05-0.5 mcg/kg/min. The treating physician may alter the target mean arterial pressure if clinically indicated.
  Arms: Norepinephrine and vasopressin
Drug: Norepinephrine — Subjects will receive norepinephrine (0.05 to 0.5 mcg/kg/min) by continuous infusion with titration by bedside nurse to achieve and maintain a target mean arterial pressure (65-75 mm Hg). The treating physician may choose the initial dosage of norepinephrine within the initial range of 0.05-0.5 mcg/kg/min. The treating physician may alter the target mean arterial pressure if clinically indicated.

SUMMARY:
Sepsis, a systemic host response to the invasion of a pathogenic microorganism, may progress to severe sepsis, wherein the patient experiences acute dysfunction in at least one organ system, and further develop into septic shock if the patient cannot regain adequate systemic blood pressure and perfusion after adequate and appropriate fluid resuscitation. Further prospective study of the potential mortality benefit with combination norepinephrine and vasopressin in critically ill patients with septic shock needs to be performed. Our research will resolve this essential question and improve the scientific knowledge surrounding vasoactive medications in patients with septic shock.

DETAILED DESCRIPTION:
Sepsis, a systemic host response to the invasion of a pathogenic microorganism, may progress to severe sepsis, wherein the patient experiences acute dysfunction in at least one organ system, and further develop into septic shock if the patient cannot regain adequate systemic blood pressure and perfusion after adequate and appropriate fluid resuscitation. The exact societal burden from severe sepsis and septic shock in difficult to quantify: millions of individuals in both industrialized and developing nations experience these syndromes each year, the best medical centers in the world have only achieved a 22% mortality rate for severe sepsis, and caregivers as well as patients endure a long-lasting impact from caring from loved ones who have survived severe sepsis. Recently, the impactful work performed by Rivers and colleagues that established early goal-directed therapy (EGDT) as the standard of care for patients with severe sepsis or septic shock has been compared to usual care in three international trials. The results of these trials suggest that usual care is as effective as EGDT, which necessitates new research be conducted into each component of EGDT to determine how and to what extent specific therapies are safe and effective. One key aspect of the provision of care to patients with septic shock is the time to initiation and choice of vasoactive agents. This study will investigate the use of norepinephrine and vasopressin versus norepinephrine alone as the initial vasoactive regimen in critically ill adult patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (no maximum age)
* At least 2 of 4 systemic inflammatory response syndrome criteria:

  1. Fever (>38°C) or hypothermia (<36°C),
  2. Tachycardia (heart rate >90 bpm),
  3. Tachypnea (respiratory rate >20 breaths/min or partial pressure of carbon dioxide <4.3 kPa) or need for mechanical ventilation,
  4. Abnormal leucocyte count (>12000 cells/mm3, <4000 cells/mm3 or >10% immature (band) forms).
* Hypotension despite adequate intravenous fluid resuscitation (minimum 20 mL/kg within the previous 4 hours)
* Clinical suspicion for or confirmation of an infection
* Admitted or being admitted to the medical intensive care unit

Exclusion Criteria:

* End-stage renal disease requiring long-term dialysis
* Pregnant
* Not expected to be alive within 48 hours of enrollment
* Receipt of a continuous infusion of vasoactive medication(s) other than use for emergency stabilization of blood pressure (for less than 4 hours)
* Enrollment in another clinical trial within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Time to goal MAP | Within 28 days of therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Drayton Hammond, Pharm.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hammond DA, Ficek OA, Painter JT, McCain K, Cullen J, Brotherton AL, Kakkera K, Chopra D, Meena N. Prospective Open-label Trial of Early Concomitant Vasopressin and Norepinephrine Therapy versus Initial Norepinephrine Monotherapy in Septic Shock. Pharmacotherapy. 2018 May;38(5):531-538. doi: 10.1002/phar.2105. Epub 2018 Apr 30. PMID 29600824